CLINICAL TRIAL: NCT02936102
Title: A Phase I, Open-label, Multi-center Dose Escalation Study of FAZ053 as Single Agent and in Combination With PDR001 in Adult Patients With Advanced Malignancies
Brief Title: A Study of FAZ053 Single Agent and in Combination With PDR001 in Patients With Advanced Malignancies.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The early termination was based on a business decision that FAZ053 would no longer be formulated and was not a consequence of any safety concern.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFAZ053X2101; 2016-001470-15 (EudraCT Number)
Record Dates: First submitted 2016-09-15; First posted 2016-10-18 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors; Triple Negative Breast Cancer; Chordoma and Alveolar Soft Part Sarcoma
Keywords: Phase I; FAZ053; PDR001; Checkpoint inhibitor; PD-L1; PD-1
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Chordoma; Sarcoma, Alveolar Soft Part | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FAZ053 single agent (Experimental)
  Interventions: Drug: FAZ053
- FAZ053 + PDR001 (Experimental)
  Interventions: Drug: FAZ053; Drug: PDR001

INTERVENTIONS:
Drug: FAZ053 — Anti-PD-L1 Antibody
Drug: PDR001 — Anti-PD-1 Antibody
  Arms: FAZ053 + PDR001

SUMMARY:
The purpose of this "first-in-human" study of FAZ053 is to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and antitumor activity of FAZ053 administered Intravenously (i.v.)as a single agent or in combination with PDR001 in adult patients with advanced solid tumors.

By blocking the interaction between Programmed Death Ligand-1 (PD-L1) and its receptors, Programmed Death-1 (PD-1) and B7.1, FAZ053 inhibits the PD-L1 immune checkpoint, resulting in activation of an antitumor immune response by activating effector T-cells and inhibiting regulatory T-cells.

This study has been designed as a Phase I, open-label, multi-center study with a dose escalation part of FAZ053 as single agent and in combination with PDR001, followed by a dose expansion part of FAZ053 as single agent.

FAZ053 will initially be dosed every three weeks. A less frequent dosing regimen such as every 6 weeks may be evaluated in parallel.

A patient may continue treatment with FAZ053 single agent or in combination with PDR001 until the patient experiences unacceptable toxicity, confirmed disease progression per immune related Response Criteria and/or treatment is discontinued at the discretion of the investigator or the patient.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any procedure.
* Dose escalation cohorts of FAZ053 single agent and FAZ053 in combination with PDR001: Patients with advanced/metastatic solid tumors with measurable or non-measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 who may or may not have received prior treatment with an immune checkpoint inhibitor, who have progressed despite standard therapy, or for whom no standard therapy is available.
* Dose expansion groups of FAZ053 single agent: Patients with advanced/metastatic solid tumors with at least one measurable lesion as determined by RECIST version 1.1 who may or may not have received prior treatment with an immune checkpoint inhibitor (for FAZ053 single agent no treatment with an anti-PD-L1 inhibitor is permitted), who have progressed despite standard therapy, or for whom no standard therapy is available and fit into one of the following groups:
* FAZ053 single agent: TNBC/ Chordoma/ ASPS
* Performance Status (PS) ≤ 2:
* Patient must have a site of disease amenable to biopsy and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy at screening/ baseline and during therapy on this study.

Exclusion Criteria:

* Presence of symptomatic central nervous system (CNS) metastases or CNS metastases that require local CNS-directed therapy (e.g. radiotherapy or surgery) or increasing doses of corticosteroids within the prior 2 weeks. Patients with treated brain metastases should be neurologically stable (for 4 weeks post-treatment and prior to study enrollment) and off of steroids for at least 2 weeks before administration of any study treatment.
* History of severe hypersensitivity to study treatment excipients and additives or other monoclonal antibodies (mAbs) and/or their excipients.
* Active, known or suspected autoimmune disease. Patients with vitiligo, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger should not be excluded. Patients previously exposed to anti-PD-1/PD-L1 treatment who are adequately treated for skin rash or with replacement therapy for endocrinopathies should not be excluded.
* Treatment with cytotoxic or targeted antineoplastics within 3 weeks of initiation of study treatment. For cytotoxic agents that have major delayed toxicity a washout period of one cycle is indicated (examples are nitrosoureas and mitomycin C which typically require a 6 week washout). Prior antibodies or immunotherapies require a 6 week washout.
* Patients receiving systemic chronic steroid therapy or any immunosuppressive therapy (≥ 10mg/day prednisone or equivalent). Topical, inhaled, nasal and ophthalmic steroids are allowed.
* Active infection requiring systemic antibiotic therapy.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | throughout the study and up to 150 days after end of treatment (up to approximately 46 months)
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory parameters qualifying and reported as AEs.
Incidence of Dose Limiting Toxicities (DLTs) | 21 days (single agent FAZ053) and 42 days (FAZ053+PDR001)
  A DLT is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications, which occurs within the first 21 days of treatment with FAZ053 alone or within the first 42 days when FAZ053 is given in combination with PDR001 during the dose escalation part of the study. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Dose interruptions and reductions | Up to approximately 41 months
  Number of participants with dose interruptions and reductions as a measure of tolerability.
Dose intensity | Up to approximately 41 months
  Dose intensity is defined as actual dose received divided by actual duration of exposure.

SECONDARY OUTCOMES:
Serum concentration-time profiles of FAZ053 as single agent and FAZ053 in combination with PDR001. | 41 months
Presence of anti-FAZ053 and anti-PDR001. | 41 months
Concentration of anti-FAZ053 and anti-PDR001. | 41 months
Receptor Occupancy (RO) profiles when FAZ053 is given as single agent. | 41 months
Total soluble/shed PD-L1 concentration-time profiles when FAZ053 is given as single agent and for FAZ053 in combination with PDR001. | 41 months
Histopathology of tumor infiltrating lymphocytes (TILs) by hematoxylin. | 41 months
Histopathology of tumor infiltrating lymphocytes (TILs) by eosin (H&E) stain. | 41 months
Overall response rate (ORR) per RECIST v1.1 | 41 months
Best overall response per RECIST v1.1 | 41 months
Disease control rate per RECIST 1.1 | 41 months
Progression free survival (PFS) per RECIST 1.1 | 41 months
Duration of response per RECIST 1.1 | 41 months
Overall response rate (ORR) per immune related Response Criteria (irRC). | 41 months
Progression free survival (PFS) per immune related Response Criteria (irRC). | 41 months
Characterization of Tumor Infiltrating Lymphocytes (TILs) by Immunohistochemistry (IHC) | 41 months
Characterization of myeloid cell infiltrate by IHC. | 41 months
Area under the curve (AUC) for FAZ053 as single agent and FAZ053 in combination with PDR001. | 41 months
Cmax for FAZ053 as single agent and FAZ053 in combination with PDR001. | 41 months
Tmax for FAZ053 as single agent and FAZ053 in combination with PDR001. | 41 months
Half-life for FAZ053 as single agent and FAZ053 in combination with PDR001. | 41 months
Clast for FAZ053 as single agent and FAZ053 in combination with PDR001. | 41 months
Tlast for FAZ053 as single agent and FAZ053 in combination with PDR001. | 41 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (2):
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - UT MD Anderson Cancer Center, Houston, Texas
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Toulouse, France
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Koto Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CFAZ053X2101 Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18379